CLINICAL TRIAL: NCT04844905
Title: Adjunctive Ivermectin Mass Drug Administration for Malaria Control on the Bijagos Archipelago of Guinea Bissau: A Cluster-randomized Placebo-controlled Trial
Brief Title: Adjunctive Ivermectin Mass Drug Administration for Malaria Control
Acronym: MATAMAL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Medical Research Council Unit, The Gambia (Other); Ministerio de Saude Publica, Guinee-Bissau (Unknown); Bandim Health Project (Other); Instituto Nacional de Estudos e Pesquisas, Guinee-Bissau (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19156
Record Dates: First submitted 2021-03-17; First posted 2021-04-14 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Malaria,Falciparum; Neglected Tropical Diseases; Strongyloidiasis; Lymphatic Filariasis; Scabies; Hook Worm; Soil Transmitted Helminths
Keywords: Vector Control; Mass Drug Administration; Integrated Disease Control; Malaria; Guinea Bissau; West Africa; Antimalarials; Ivermectin; Dihydroartemisinin; Piperaquine
MeSH Terms: conditions — Malaria, Falciparum; Neglected Diseases; Strongyloidiasis; Elephantiasis, Filarial; Scabies; Ancylostomiasis; Malaria | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: Two arms with clusters randomized to DP+IVM or DP+Placebo with a 1:1 ratio
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent statistician will randomize the clusters to DP+IVM or DP+Placebo. The Placebo is identical in size, shape and colour and packaging. An independent pharmacist at Medical Research Council Unit The Gambia @ London School of Hygiene and Tropical Medicine will label the IVM and Placebo according to the statistician's designation and maintain the masking from all other investigators. Specifically generated masking codes will be generated and saved in three separate encrypted locations securely. Only the statistician and the pharmacist will have access to the encryption key.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivermectin Mass Drug Administration (Experimental): Ivermectin and Dihydroartemisinin-piperaquine MDA will be given to all eligible participants in each cluster (island) in addition to the standard national malaria control programme interventions.
  Interventions: Drug: Ivermectin; Drug: Dihydroartemisinin-piperaquine
- Placebo Mass Drug Administration (Placebo Comparator): Placebo and Dihydroartemisinin-piperaquine MDA will be given to all eligible participants in each cluster (island) in addition to the standard national malaria control programme interventions.
  Interventions: Drug: Placebo; Drug: Dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: Ivermectin — Ivermectin will be given as tablets of 3 or 6mg. It will be given at 300-400μg/kg/day for 3 days (to the nearest whole tablet) each month for 3 months. It will be taken on an empty stomach with water.
  Arms: Ivermectin Mass Drug Administration
Drug: Placebo — Placebo will be given as tablets of 3 or 6mg (identical to Ivermectin in colour, size, shape and packaging). It will be given at 300-400μg/kg/day for 3 days (to the nearest whole tablet) each month for 3 months. It will be taken by mouth with water and without food.
  Arms: Placebo Mass Drug Administration
Drug: Dihydroartemisinin-piperaquine — Dihydroartemisinin-piperaquine will be given as tablets of 320/40mg (adult) and 160/20mg (child) piperaquine/dihydroartemisinin per tablet. Administration of a full course of dihydroartemisinin-piperaquine will be given in accordance with the manufacturer's guidelines once daily for 3 days each month for 3 months according to body weight. Dihydroartemisinin-piperaquine will be taken by mouth with water and without food.
  Other Names: Eurartesim

SUMMARY:
This is a cluster-randomized placebo-controlled clinical trial to evaluate the additive benefit of Ivermectin (IVM) (or Placebo) mass drug administration (MDA) to dihydroartemisinin-piperaquine (DP) MDA for malaria control in a moderate to low malaria-endemic setting as an adjunctive strategy to existing programmatic malaria control measures. The regime of DP and IVM will target both human reservoirs of Plasmodium falciparum and the Anopheles gambiae vector respectively, with the aim of interrupting transmission. The trial will be conducted on the Bijagos Archipelago, where islands (clusters) will be randomised to receive seasonal DP and IVM or DP and Placebo MDA. The primary outcome will be the prevalence of infection with Plasmodium falciparum in all age groups detected by nucleic acid amplification testing during the peak malaria transmission season after two years of intervention.

DETAILED DESCRIPTION:
The objectives of this trial are

1. To evaluate the impact of adjunctive IVM to DP MDA on malaria transmission in communities with high ITN coverage.
2. To evaluate the impact of IVM MDA on An. gambiae population density and age-structure.
3. To evaluate the impact of IVM MDA on the prevalence of co-endemic IVM-susceptible Neglected Tropical Diseases (lymphatic filariasis, soil transmitted helminths and scabies)
4. To evaluate acceptability, feasibility and access to MDA as a strategy for malaria control and to identify the most acceptable way of achieving and sustaining high coverage MDA with IVM and DP.

This cluster-randomized placebo-controlled trial has two arms. A total of 24 clusters will be randomly assigned to receive DP + IVM MDA or DP+ Placebo MDA using computer-generated random numbers. To mitigate against contamination effects, the majority of clusters will be separate islands and will be separated by distances greater than 2km. On the two islands that are divided (each into two clusters), a buffer zone of 2km between each cluster will be ensured. The total population of the archipelago is 24,000. The investigators will ensure balance between trial arms with respect to population size, baseline Plasmodium falciparum prevalence and access to health care. All clusters will receive the standard programmatic malaria control interventions implemented by the National Malaria Control Programme which includes insecticide-treated nets (ITN), intermittent preventative treatment in pregnancy (IPTp), seasonal malarial chemoprophylaxis (SMC) for children aged 3-59 months and case diagnosis and treatment (CDT) with Artemether-lumefantrine.

ELIGIBILITY:
Inclusion Criteria:

1. Age over six months to receive dihydroartemisinin-piperaquine
2. Height over 90cm or weight over 15kg to receive ivermectin or placebo
3. Willingness to adhere to trial procedures
4. Individual written, informed consent from the participant or parent/guardian in the case of participants below the age of 18 years (and assent in young people between the ages of 12 and 17 years of age)

Exclusion Criteria:

1. Known severe chronic illness (AIDS, Tuberculosis, chronic malnutrition)
2. Known hypersensitivity to either dihydroartemisinin-piperaquine or ivermectin
3. Pregnancy (any trimester) and breastfeeding (for ivermectin (or placebo)) and pregnancy (first trimester only) (for dihydroartemisinin-piperaquine)
4. Travel to a Loa loa endemic country (eg Central African Republic) (for ivermectin (or placebo))
5. Concomitant drugs that influence cardiac function or affect the corrected QT interval (for dihydroartemisinin-piperaquine)

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24000 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence of infection with Plasmodium falciparum | 2 years
  Prevalence of infection with Plasmodium falciparum in all age groups estimated using a cross-sectional survey sample conducted during peak transmission season after 2 years of intervention

SECONDARY OUTCOMES:
Vector parous rate | 7-14 days post-MDA
  Vector parous rate will be determined by assessment of mosquitoes trapped 7-14 days following MDA. Vector parity will be used to determine Anopheles gambiae age structure to estimate vector survival between arms.
Prevalence of infection with Plasmodium falciparum | 1 year
  Prevalence of infection with Plasmodium falciparum in all age groups estimated using a cross-sectional survey sample conducted after the first year of intervention
Incidence of clinical malaria (Passive Case Detection) | For six months during the malaria transmission season
  Incidence of clinical malaria diagnosed at health facilities confirmed by malaria Rapid Diagnostic Test
Incidence of clinical malaria (Active Case Detection) | For six months during the malaria transmission season
  Incidence of clinical malaria confirmed by malaria Rapid Diagnostic Test in a cohort of 50 children per cluster aged 5-14 years
Age-adjusted prevalence of recent exposure to Plasmodium falciparum | Peak transmission season at 1 year and 2 years
  Mean Median Fluorescence Intensity of serological markers associated with recent exposure to Plasmodium falciparum in all age groups estimated using a cross-sectional survey sample during peak transmission season after each year of intervention
Vector density | For six months during the malaria transmission season
  Total number of trapped mosquitoes per cluster
Vector species composition | For six months during the malaria transmission season
  Species characterisation using nucleic acid amplification tests as a proportion of total mosquitoes caught in traps
Prevalence of exposure to Anopheles exposure | Peak transmission season at 1 year and 2 years
  Mean Median Fluorescence Intensity of serological markers associated with exposure to Anopheles salivary antigen in all age groups estimated using a cross-sectional survey sample
Vector sporozoite rates | For six months during the malaria transmission season
  Proportion of Plasmodium falciparum circumsporozoite antibody (CSP) positive mosquitoes caught in traps
Prevalence of Ivermectin-susceptible Neglected Tropical Diseases (NTDs) | 2 years
  Prevalence of IVM-susceptible NTDs (scabies, strongyloides, other soil-transmitted helminths and lymphatic filariasis) and head lice using clinical and serological parameters estimated using a cross-sectional survey sample during the dry season after two years of intervention.
MDA coverage estimates | During MDA in year 1 and year 2
  Cluster level coverage estimates calculated from MDA distribution and denominator census
Prevalence of resistance to artemisinin and partner drugs in humans | Peak transmission season at 1 year and at 2 years
  Prevalence of resistance to artemisinin and partner drugs in humans using molecular markers of resistance in all age groups estimated using a cross-sectional survey sample

CONTACTS AND LOCATIONS:
Overall Officials: Anna R Last, MBChB PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Bijagos Archipelago (islands), Bissau, Guinea-Bissau

IPD SHARING:
Plan to Share IPD: Yes
There is a manuscript in preparation detailing the study protocol and statistical analysis plan. The participant information and and informed consent form may be requested from the trial research team. Results and a clinical study report will be made available within six months of completion of the trial. Analytic code will be made available under a Creative Commons license. Publication of results will be open-access and available in pre-print on MedRxiv (The Preprint Server for Health Sciences).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The study protocol and Statistical Analysis Plan (SAP) will be made available on acceptance of the manuscript for publication. Participant information and Informed Consent Form (ICF) will be made available from recruitment. Results (including Clinical Study Report (CSR)) will be made available within six months of completion of the trial.
Access Criteria: Study Protocol and Statistical Analysis Plan (SAP) will be published in an Open Access peer-reviewed journal. The participant information and and informed consent form may be requested from the trial research team. Results and a clinical study report will be made available within six months of completion of the trial. Analytic code will be made available under a Creative Commons license. Publication of results will be Open-Access and available in pre-print on MedRxiv (The Preprint Server for Health Sciences).

REFERENCES:
- [Derived] Hutchins H, Pretorius E, Bradley J, Teixeira da Silva E, Vasileva H, Ndiath MO, Jones RT, Soumare HDM, Nyang H, Prom A, Sambou S, Ceesay F, Ceesay S, Moss S, Mabey D, Djata P, Nante JE, Martins C, Logan JG, Slater H, Tetteh K, Drakeley C, D'Alessandro U, Rodrigues A, Last A. Adjunctive ivermectin mass drug administration for malaria control on the Bijagos Archipelago of Guinea-Bissau (MATAMAL): a quadruple-blinded, cluster-randomised, placebo-controlled trial. Lancet Infect Dis. 2025 Apr;25(4):424-434. doi: 10.1016/S1473-3099(24)00580-2. Epub 2024 Nov 14. PMID 39551062
- [Derived] Hutchins H, Bradley J, Pretorius E, Teixeira da Silva E, Vasileva H, Jones RT, Ndiath MO, Dit Massire Soumare H, Mabey D, Nante EJ, Martins C, Logan JG, Slater H, Drakeley C, D'Alessandro U, Rodrigues A, Last AR. Protocol for a cluster randomised placebo-controlled trial of adjunctive ivermectin mass drug administration for malaria control on the Bijagos Archipelago of Guinea-Bissau: the MATAMAL trial. BMJ Open. 2023 Jul 7;13(7):e072347. doi: 10.1136/bmjopen-2023-072347. PMID 37419638